CLINICAL TRIAL: NCT04212689
Title: The Effectiveness of Game-Based Virtual Reality Approach in Patients With Multiple Sclerosis
Brief Title: Virtual Reality Approach in Multiple Sclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 31.10.2019/104
Record Dates: First submitted 2019-12-25; First posted 2019-12-27 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Rehabilitation; Multiple Sclerosis
Keywords: Rehabilitation; Physiotherapy and Rehabilitation; Virtual Reality; Multiple Sclerosis; Upper extremity
MeSH Terms: conditions — Multiple Sclerosis | interventions — Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Number of participants in this group is anticipated to be 20. Conventional physiotherapy and rehabilitation methods will be applied to this group. Physiotherapy approaches include stretching exercises, neurodevelopmental approaches, static positioning, strengthening exercises, Transcutaneous Electrical Nerve Stimulation (TENS), hydrotherapy, cryotherapy.
  Interventions: Other: Conventional Physiotherapy and Rehabilitation
- Study Group (Active Comparator): Number of participants in this group is anticipated to be 20. Participants in this group will be receiving conventional physiotherapy and rehabilitation methods and 10 minutes of exercise with the game-based virtual reality system (USE-IT). In the USE-IT system two games will be played for 5 minutes each.
  Interventions: Device: Game Based Virtual Reality Exercises; Other: Conventional Physiotherapy and Rehabilitation

INTERVENTIONS:
Device: Game Based Virtual Reality Exercises — A game-based virtual reality device named USE-IT will be added to the rehabilitation program. USE-IT is a technological rehabilitation system designed by the Department of Physiotherapy and Rehabilitation at Hacettepe University. It is a smart gaming device which has been used in patients who suffer from movement loss in their upper extremities due to various neurological and orthopedic reasons.
  Arms: Study Group
Other: Conventional Physiotherapy and Rehabilitation — The conventional physiotherapy and rehabilitation program includes stretching exercises, neurodevelopmental approaches, static positioning, strengthening exercises, Transcutaneous Electrical Nerve Stimulation (TENS), hydrotherapy, cryotherapy.

SUMMARY:
The aim of our study is to investigate the effects of game-based virtual reality exercise added to conventional physiotherapy and rehabilitation program in patients with Multiple Sclerosis (MS). In order to evaluate its effectiveness, assessment of pain, range of motion and disability will be applied.

DETAILED DESCRIPTION:
Multiple Sclerosis (MS) is a neuromuscular disease that causes various degrees of disability in mobility and functional activities, causing restrictions on the individual's social and professional life, creating advanced disability and impairing quality of life. Problems in upper limb function affect quality of life and functional independence of the patients. Recovery of restricted daily life functions (such as dressing, personal care, eating and body care) is one of the main goals of physiotherapy and rehabilitation in MS and currently, conventional physiotherapy and rehabilitation methods are most commonly used. The main purpose of this method is to reduce pain, increase range of motion and muscle strength. With the developing technology various virtual reality applications have begun to take place in physiotherapy and rehabilitation programs recently. These virtual reality applications are used to motivate the patient and keep their interest in the rehabilitation. The aim of our study is to investigate the effects of game-based virtual reality exercises added to conventional physiotherapy and rehabilitation program in patients with MS.

ELIGIBILITY:
Inclusion Criteria:

* Volunteered to participate in the study,
* Aged 18-65 years
* Having a score between 1.5 - 7 according to Expanded Disability Status Scale (EDSS)

Exclusion Criteria:

* Any visual or hearing problem,
* Other neurological, orthopedic or rheumatic problems that may restrict shoulder motion or cause pain,
* Having a physical disability or uncontrolled chronic systemic disease,
* Major trauma,
* Treatment for shoulder problems within the last 6 months,
* History of epileptic attacks
* Not being stable for MS attacks during the last 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-01-20 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in range of motion from baseline to week 4 | 4 weeks
  The range of motion of the joints in the upper extremities will be measured using the universal goniometer before and after the treatment.
Change in level of pain from baseline to week 4 | 4 weeks
  Level of Pain will be assessed with Visual Analogue Scale (VAS). It is widely used among the methods of measuring the severity of pain. Scale is a 10 cm ruler, participants will mark the level of pain between 0-10 cm, 0 would means ''no pain'' and 10 would means ''worst possible pain''.
Change in disability of the upper extremity from baseline to week 4 | 4 weeks
  Disability of the upper extremities will be assessed with 'The Disabilities of the Arm, Shoulder and Hand (DASH) Questionnaire'. It is a self-administered region-specific outcome instrument developed as a measure of self-rated upper-extremity disability and symptoms. The questionnaire was designed to help describe the disability experienced by people with upper-limb disorders and also to monitor changes in symptoms and function over time.
Change in pain threshold from baseline to week 4 | 4 weeks
  The pain threshold will be measured with a digital algometer device. Algometers are devices that can be used to identify the pressure and/or force eliciting a pressure-pain threshold. It has been noted in pressure-pain threshold studies that the rate at which manual force is applied should be consistent to provide the greatest reliability.
Change in proprioception from baseline to week 4 | 4 weeks
  Proprioception will be evaluated with 'Marmara Visual Auditory Joint Education Device (MarVAJED) which was developed by the Faculty of Health Sciences of Marmara University, Istanbul. This device evaluates motion deficits of joints, analyzes joint position sense, provides biofeedback support to increase joint control and also directs to controlled exercises. It analyzes the motion of the joint with the help of small sensors and transfers the data obtained to the mobile phone, tablet or computer.
Change in kinesiophobia from baseline to week 4 | 4 weeks
  In the assessment of kinesiophobia 'Tampa Kinesiophobia Scale (TKS)' will be used. It is a 17 item questionnaire used to assess the subjective rating of kinesiophobia or fear of movement. The scale is based on the model of fear avoidance, fear of work related activities, fear of movement and fear of re-injury.
Satisfaction of the Treatment | 4 weeks
  An objective test that evaluates the satisfaction of the patient from pain status, functionality, treatment and physiotherapist after treatment will be assessed with 4 questions, and each question is given a score of 0-10 using the VAS scale. 0 means ''I am not satisfied at all'', 10 means ''I am very satisfied''.
Change in muscle strength from baseline to week 4 | 4 weeks
  The muscle strength of shoulder flexion, abduction, adduction, external and internal rotation movements will be evaluated by using the Baseline Push-Pull (New York) dynamometer. Results will be calculated in kg (1 lb = 0.454 kg). The patient's arm will be stabilized and the patient will be asked to show maximum resistance within 2 sec against the dynamometer placed and then hold it for 5 seconds at this position and power. The measurement will be repeated twice and recorded with the average of these two values.
Change in disability of the fingers from baseline to week 4 | 4 weeks
  The Nine-Hole Peg Test (9HPT) will be used to measure finger dexterity. The test is administered by asking the client to take the pegs from a container, one by one, and place them into the holes on the board, as quickly as possible. Participants must then remove the pegs from the holes, one by one, and replace them back into the container. Scores are based on the time taken to complete the test activity, recorded in seconds.
Change in spasticity from baseline to week 4 | 4 weeks
  Spasticity will be defined with Modified Ashworth Scale (MAS). The MAS measures resistance during passive soft-tissue stretching. Scoring: 0= normal tone. 1= slight increase in muscle tone, minimal resistance at the end of the range of motion (ROM) when the affected part(s) is moved in flexion or extension. 1+= slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder of the ROM. 2= more marked increase in muscle tone through most of the ROM, but affected part(s) easily moved. 3= considerable increase in muscle tone, passive movement difficult. 4= affected part(s) rigid in flexion or extension.

CONTACTS AND LOCATIONS:
Overall Officials: Nimet Sermenli Aydın, MSc, Principal Investigator — Marmara University Institute of Health Sciences; Dilara Merve Sari, MSc, Principal Investigator — Marmara University Institute of Health Sciences; Zubeyir Sari, Assoc Prof, Study Director — Marmara University Faculty of Health Sciences
Locations (1):
- Cadde Tıp Merkezi - Cadde Medical Center, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bao X, Mao Y, Lin Q, Qiu Y, Chen S, Li L, Cates RS, Zhou S, Huang D. Mechanism of Kinect-based virtual reality training for motor functional recovery of upper limbs after subacute stroke. Neural Regen Res. 2013 Nov 5;8(31):2904-13. doi: 10.3969/j.issn.1673-5374.2013.31.003. PMID 25206611
- [Background] Arman N, Tarakci E, Tarakci D, Kasapcopur O. Effects of Video Games-Based Task-Oriented Activity Training (Xbox 360 Kinect) on Activity Performance and Participation in Patients With Juvenile Idiopathic Arthritis: A Randomized Clinical Trial. Am J Phys Med Rehabil. 2019 Mar;98(3):174-181. doi: 10.1097/PHM.0000000000001001. PMID 30020092
- [Background] Burdea GC. Virtual rehabilitation--benefits and challenges. Methods Inf Med. 2003;42(5):519-23. PMID 14654886
- [Background] Rubin BD, Kibler WB. Fundamental principles of shoulder rehabilitation: conservative to postoperative management. Arthroscopy. 2002 Nov-Dec;18(9 Suppl 2):29-39. doi: 10.1053/jars.2002.36507. No abstract available. PMID 12426529
- [Background] Chen CC. Multimedia virtualized environment for shoulder pain rehabilitation. J Phys Ther Sci. 2016 Apr;28(4):1349-54. doi: 10.1589/jpts.28.1349. Epub 2016 Apr 28. PMID 27190481
- [Background] Andrews AW, Thomas MW, Bohannon RW. Normative values for isometric muscle force measurements obtained with hand-held dynamometers. Phys Ther. 1996 Mar;76(3):248-59. doi: 10.1093/ptj/76.3.248. PMID 8602410
- [Background] Bjartmar C, Trapp BD. Axonal and neuronal degeneration in multiple sclerosis: mechanisms and functional consequences. Curr Opin Neurol. 2001 Jun;14(3):271-8. doi: 10.1097/00019052-200106000-00003. PMID 11371748
- [Background] Crayton H, Heyman RA, Rossman HS. A multimodal approach to managing the symptoms of multiple sclerosis. Neurology. 2004 Dec 14;63(11 Suppl 5):S12-8. doi: 10.1212/wnl.63.11_suppl_5.s12. PMID 15596731
- [Background] Earhart GM, Cavanaugh JT, Ellis T, Ford MP, Foreman KB, Dibble L. The 9-hole PEG test of upper extremity function: average values, test-retest reliability, and factors contributing to performance in people with Parkinson disease. J Neurol Phys Ther. 2011 Dec;35(4):157-63. doi: 10.1097/NPT.0b013e318235da08. PMID 22020457
- [Background] Feys P, Helsen W, Liu X, Mooren D, Albrecht H, Nuttin B, Ketelaer P. Effects of peripheral cooling on intention tremor in multiple sclerosis. J Neurol Neurosurg Psychiatry. 2005 Mar;76(3):373-9. doi: 10.1136/jnnp.2004.044305. PMID 15716530
- [Background] Hiller LB, Wade CK. Upper extremity functional assessment scales in children with Duchenne muscular dystrophy: a comparison. Arch Phys Med Rehabil. 1992 Jun;73(6):527-34. PMID 1622300
- [Background] Peresedova AV, Chernikova LA, Zavalishin IA. [Physical rehabilitation in multiple sclerosis: general principles and high-tech approaches]. Vestn Ross Akad Med Nauk. 2013;(10):14-21. Russian. PMID 24640715